CLINICAL TRIAL: NCT01121588
Title: PHASE 1B OPEN-LABEL STUDY OF THE SAFETY AND CLINICAL ACTIVITY OF CRIZOTINIB (PF-02341066) IN TUMORS WITH GENETIC EVENTS INVOLVING THE ANAPLASTIC LYMPHOMA KINASE (ALK ) GENE LOCUS
Brief Title: Studying An Investigational Drug Crizotinib (PF-02341066) In Non Non-Small Cell Lung Cancer Tumors That Are Positive For Anaplastic Lymphoma Kinase (ALK)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Termination of further treatment on the study due to the availability of commercial supply or a rollover study (NCT05160922) that will allow active subjects to continue receiving treatment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8081013; 2010-022978-14 (EudraCT Number)
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Neoplasms Malignant
Keywords: neoplasm malignant; lymphoma; neuroblastoma; Crizotinib; anaplastic lymphoma kinase; ALK
MeSH Terms: conditions — Neoplasms; Lymphoma; Neuroblastoma | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Crizotinib (Experimental)
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Crizotinib tablets, 250 mg BID, will be administered orally on a continuous dosing schedule
  Other Names: PF-02341066

SUMMARY:
This is a Phase 1 trial evaluating the safety and efficacy of crizotinib in patients with tumors except non-small cell lung cancer that are positive for ALK.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven diagnosis of malignancy other than NSCLC
* positive for translocation or inversion event involving the ALK gene locus
* positive for ALK amplification events
* positive for ALK activating point mutations

Exclusion Criteria:

* mutations of amplifications involving the c-Met gene but not the ALK gene
* concurrent treatment on another therapeutic clinical trial
* prior therapy specifically directed against ALK

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03-22 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (9):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highland Oncology Group, Springdale, Arkansas
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OHSU Center for Health and Healing 2, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Greenville Health System, Institute for Translational Oncology Research, Greenville, South Carolina
- China (2):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Chaoyang District
  - SUN Yat-Sen University Cancer Center, Guangzhou, Guangdong
- Italy (2):
  - Centro di Ricerca di Fase 1 ASST-Monza, Monza
  - PO San Gerardo, ASST Monza-U.O Ematologia, Monza
- Japan (3):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
- Russia (2):
  - GBOU VPO "First Saint-Petersburg State Medical University n.a.I.P Pavlov" Ministry of Health, Saint Petersburg
  - Institute of Pedriatric Oncology, Hematology and Transplantation n.a R.M Gorbacheva, Saint Petersburg
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- National Taiwan University Hospital, Department of Internal Medicine, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081013&StudyName=An%20Investigational%20Drug%2C%20Crizotinib%20%28PF-02341066%29%2C%20Is%20Being%20Studied%20In%20Tumors%2C%20Except%20Non-Small%20Cell%20Lung%20Cancer%2C%20That%20Are%20Posit

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 44 Anaplastic lymphoma kinase (ALK) genetic event positive participants were enrolled into the study and treated: 17 with anaplastic large cell lymphoma (ALCL), 9 with inflammatory myofibroblastic tumors (IMT), and 18 with other tumors (ALK-positive malignancies excluding non-small cell lung cancer).
Groups:
- ALCL Arm: In ALK genetic event positive participants with ALCL, crizotinib 250 mg twice daily (BID) was administered orally at approximately the same time each day on a continuous daily dosing schedule. Crizotinib was allowed to be taken without regard to meals. Cycles were defined in 21 day periods. Participants could have continued treatment with crizotinib on this study as long as there was evidence of clinical benefit in the judgment of the Investigator.
- IMT Arm: In ALK genetic event positive participants with IMT, crizotinib 250 mg twice daily (BID) was administered orally at approximately the same time each day on a continuous daily dosing schedule. Crizotinib was allowed to be taken without regard to meals. Cycles were defined in 21 day periods. Participants could have continued treatment with crizotinib on this study as long as there was evidence of clinical benefit in the judgment of the Investigator.
- Other Tumors: In ALK genetic event positive participants with other tumors (excluding non-small cell lung cancer), crizotinib 250 mg twice daily (BID) was administered orally at approximately the same time each day on a continuous daily dosing schedule. Crizotinib was allowed to be taken without regard to meals. Cycles were defined in 21 day periods. Participants could have continued treatment with crizotinib on this study as long as there was evidence of clinical benefit in the judgment of the Investigator.
Period: Overall Study
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Started | 17 | 9 | 18
Completed | 0 | 0 | 0
Not Completed | 17 | 9 | 18
Not completed — Death | 5 | 3 | 13
Not completed — Study Terminated by Sponsor | 1 | 1 | 0
Not completed — Participant Refused Further Followup | 2 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Non-Specified Reasons | 9 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Baseline population included all enrolled participants who received at least one dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | ALCL Arm | IMT Arm | Other Tumors | Total
Number analyzed (Participants) | 17 | 9 | 18 | 44
Age, Continuous [Median (Full Range); unit: Years] — Population: The data for age was provided for the overall population and the pediatric population. Number Analyzed for Overall Population = Number of participants (regardless of age) with the corresponding type(s) of tumor, who were enrolled and treated in this study. Number Analyzed for Pediatric Population = Number of participants <18 years of age with the corresponding type(s) of tumor, who were enrolled and treated in this study.
  Years
    Overall Population | 25.0 [15.0 to 37.0] | 32.0 [16.0 to 73.0] | 49.0 [18.0 to 73.0] | 32.0 [15.0 to 73.0]
    Pediatric Population: number analyzed (Participants) | 3 | 2 | 0 | 5
    Pediatric Population | 15.0 [15.0 to 16.0] | 16.5 [16.0 to 17.0] |  | 16.0 [15.0 to 17.0]
Age, Customized [Count of Participants; unit: Participants] — Number Analyzed for Overall Population = Number of participants (regardless of age) with the corresponding type(s) of tumor, who were enrolled and treated in this study.
  Participants
    <18 | 3 | 2 | 0 | 5
    Between 18 and 65 years | 14 | 6 | 15 | 35
    >=65 years | 0 | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The data for sex was provided for the overall population and the pediatric population. Number Analyzed for Overall Population = Number of participants (regardless of age) with the corresponding type(s) of tumor, who were enrolled and treated in this study. Number Analyzed for Pediatric Population = Number of participants <18 years of age with the corresponding type(s) of tumor, who were enrolled and treated in this study.
  Participants
    Overall population: Female | 5 | 4 | 10 | 19
    Overall population: Male | 12 | 5 | 8 | 25
    Pediatric Population: number analyzed (Participants) | 3 | 2 | 0 | 5
    Pediatric Population: Female | 1 | 1 | 0 | 2
    Pediatric Population: Male | 2 | 1 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 4 | 7 | 23
  Black | 0 | 0 | 0 | 0
  Asian | 5 | 5 | 11 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Racial Designation for pediatric population. Population: Number Analyzed for Pediatric Population = Number of participants <18 years of age with the corresponding type(s) of tumor, who were enrolled and treated in this study.
  Participants
    White: number analyzed (Participants) | 3 | 2 | 0 | 5
    White | 1 | 0 | 0 | 1
    Black: number analyzed (Participants) | 3 | 2 | 0 | 5
    Black | 0 | 0 | 0 | 0
    Asia: number analyzed (Participants) | 3 | 2 | 0 | 5
    Asia | 2 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-Causality Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Serious AE was an AE resulting in death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity, congenital anomaly. Treatment-emergent AEs were those with initial onset or that worsened in severity after the first dose of study medication. Grades of AEs were defined by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 4.03. Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care activity of daily living (ADL); Grade 4=events with life-threatening consequences, urgent intervention indicated; Grade 5=death related to AE.
Time Frame: From the first dose of study treatment up to 28 days after the last dose of study treatment (maximum 444 weeks)
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 17 | 9 | 18
Participants
  AEs | 17 | 9 | 17
  SAEs | 8 | 4 | 7
  Maximum Grade 3 or 4 AEs | 13 | 7 | 8
  Maximum Grade 5 AEs | 2 | 0 | 4
  AEs resulting in study treatment discontinuation (participant continued study) | 1 | 0 | 3
  AEs resulting in dose reduction | 4 | 1 | 3
  AEs resulting in temporary discontinuation of study treatment | 8 | 6 | 10

2. Primary Outcome: Number of Participants With All-Causality TEAEs in the Pediatric Population
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Serious AE was an AE resulting in death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity, congenital anomaly. Treatment-emergent AEs were those with initial onset or that worsened in severity after the first dose of study medication.Grades of AEs were defined by NCI CTCAE version 4.03. Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4=events with life-threatening consequences, urgent intervention indicated; Grade 5=death related to AE.
Time Frame: From the first dose of study treatment up to 28 days after the last dose of study treatment (maximum 342 weeks)
Population: Enrolled pediatric (<18 years old) participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 3 | 2 | 0
Participants
  AEs | 3 | 2 |
  SAEs | 2 | 1 |
  Maximum Grade 3 or 4 AEs | 3 | 2 |
  Maximum Grade 5 AEs | 0 | 0 |
  AEs resulting in study treatment discontinuation (participant continued study) | 0 | 0 |
  AEs resulting in dose reduction | 1 | 0 |
  AEs resulting in temporary discontinuation of study treatment | 2 | 2 |

3. Primary Outcome: Number of Participants With Treatment-Related TEAEs
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were those with initial onset or that worsened in severity after the first dose of study medication. Grades of AEs were defined by NCI CTCAE version 4.03. Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4=events with life-threatening consequences, urgent intervention indicated; Grade 5=death related to AE.
Time Frame: From the first dose of study treatment up to 28 days after the last dose of study treatment (maximum 444 weeks)
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 17 | 9 | 18
Participants
  AEs | 16 | 8 | 15
  SAEs | 5 | 3 | 2
  Maximum Grade 3 or 4 AEs | 11 | 5 | 6
  Maximum Grade 5 AEs | 0 | 0 | 2
  AEs resulting in study treatment discontinuation (participant continued study treatment) | 0 | 0 | 2
  AEs resulting in dose reduction | 4 | 1 | 3
  AEs resulting in temporary discontinuation of study treatment | 6 | 4 | 6

4. Primary Outcome: Number of Participants With Treatment-Related TEAEs in the Pediatric Population
Description: as for outcome 3
Time Frame: From the first dose of study treatment up to 28 days after the last dose of study treatment (maximum 342 weeks)
Population: Enrolled pediatric (<18 years old) participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 3 | 2 | 0
Participants
  AEs | 3 | 2 |
  SAEs | 2 | 1 |
  Maximum Grade 3 or 4 AEs | 2 | 1 |
  Maximum Grade 5 AEs | 0 | 0 |
  AEs resulting in study treatment discontinuation (participant continued study treatment) | 0 | 0 |
  AEs resulting in dose reduction | 1 | 0 |
  AEs resulting in temporary discontinuation of study treatment | 1 | 1 |

5. Primary Outcome: Number of Participants With Laboratory Test Results Shifted From Grade <=2 At Baseline to Grade 3 or 4 Postbaseline (Hematology and Chemistries)
Description: Baseline assessment was defined as the last assessment performed on or prior to the date of the first dose of study treatment. Both hematology and clinical chemistry parameters were analyzed. Grades of severity were defined by CTCAE v4.0. Grade 1 = mild adverse event; Grade 2 = moderate adverse event; Grade 3= severe adverse event; Grade 4 = life-threatening consequences; urgent intervention indicated.
Time Frame: From the first dose of study treatment up to 28 days after the last dose of study treatment (maximum 444 weeks)
Population: Number analyzed = Number of participants with a postbaseline value during the study treatment for this outcome measure for each specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 16 | 9 | 16
Participants
  Anemia | 1 | 0 | 5
  Hemoglobin increased | 0 | 0 | 0
  Lymphocyte count decreased | 1 | 1 | 4
  Lymphocyte count increased | 0 | 0 | 0
  Neutrophil count decreased | 8 | 3 | 1
  Platelet count decreased | 0 | 0 | 0
  White blood cell decreased | 3 | 0 | 1
  Alanine aminotransferase increased | 2 | 1 | 2
  Alkaline phosphatase increased | 0 | 0 | 0
  Aspartate aminotransferase increased | 4 | 0 | 1
  Blood bilirubin increased | 0 | 0 | 1
  Creatinine increased | 0 | 0 | 0
  Hypercalcemia: number analyzed (Participants) | 16 | 9 | 14
  Hypercalcemia | 0 | 0 | 0
  Hyperglycemia | 0 | 0 | 0
  Hyperkalemia | 2 | 0 | 0
  Hypermagnesemia: number analyzed (Participants) | 16 | 9 | 14
  Hypermagnesemia | 0 | 0 | 1
  Hypernatremia | 0 | 0 | 0
  Hypoalbuminemia | 0 | 0 | 2
  Hypocalcemia: number analyzed (Participants) | 16 | 9 | 14
  Hypocalcemia | 0 | 0 | 0
  Hypoglycemia | 2 | 0 | 0
  Hypokalemia | 0 | 0 | 2
  Hypomagnesemia: number analyzed (Participants) | 16 | 9 | 14
  Hypomagnesemia | 0 | 0 | 0
  Hyponatremia | 0 | 0 | 2
  Hypophosphatemia: number analyzed (Participants) | 16 | 9 | 14
  Hypophosphatemia | 3 | 0 | 1

6. Primary Outcome: Number of Participants With Laboratory Test Results Shifted From Grade <=2 At Baseline to Grade 3 or 4 Postbaseline (Hematology and Chemistries) in the Pediatric Population
Description: Baseline assessment was defined as the last assessment performed on or prior to the date of the first dose of study treatment. Both hematology and chemistry laboratory assessments were analyzed. Grades of severity were defined by CTCAE v4.0. Grade 1 = mild adverse event; Grade 2 = moderate adverse event; Grade 3= severe adverse event; Grade 4 = life-threatening consequences; urgent intervention indicated. Unplanned laboratory test results were also included.
Time Frame: From the first dose of study treatment up to 28 days after the last dose of study treatment (maximum 342 weeks)
Population: Enrolled pediatric (<18 years old) participants who received at least 1 dose of study treatment and had both baseline and post-baseline values.
Measure: Count of Participants; unit: Participants
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 3 | 2 | 0
Participants
  Anemia | 0 | 0 | 0
  Hemoglobin increased | 0 | 0 | 0
  Lymphocyte count decreased | 1 | 0 | 0
  Lymphocyte count increased | 0 | 0 | 0
  Neutrophil count decreased | 2 | 1 | 0
  Platelet count decreased | 0 | 0 | 0
  White blood cell decreased | 2 | 0 | 0
  Alanine aminotransferase increased | 0 | 0 | 0
  Alkaline phosphatase increased | 0 | 0 | 0
  Aspartate aminotransferase increased | 1 | 0 | 0
  Blood bilirubin increased | 0 | 0 | 0
  Creatinine increased | 0 | 0 | 0
  Hypercalcemia | 0 | 0 | 0
  Hyperglycemia | 0 | 0 | 0
  Hyperkalemia | 0 | 0 | 0
  Hypermagnesemia | 0 | 0 | 0
  Hypernatremia | 0 | 0 | 0
  Hypoalbuminemia | 0 | 0 | 0
  Hypocalcemia | 0 | 0 | 0
  Hypoglycemia | 1 | 0 | 0
  Hypokalemia | 0 | 0 | 0
  Hypomagnesemia | 0 | 0 | 0
  Hyponatremia | 0 | 0 | 0
  Hypophosphatemia | 1 | 0 | 0

7. Primary Outcome: Objective Response Rate (ORR) - Percentage of Participants With Objective Response
Description: Percentage of participants with confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) (1.1) as determined by the investigators. CR = disappearance of all target lesions. PR = greater than equal to (>=) 30% decrease in sum of target lesions taking as reference baseline sum diameters. ORR based on Cheson criteria was defined similarly however, confirmation of response was not required. If participant had tumor response assessed only by RECIST or Cheson, then ORR was based on the single result. If tumor response was assessed by both RECIST and Cheson, then ORR was reported based on tumor response by Cheson criteria unless the Cheson has indeterminate result, in which case the RECIST result was reported. Participant(s) who did not have tumor assessment results from either RECIST 1.1 or Cheson criteria reported at baseline were to be excluded from the analysis.
Time Frame: From the date of first dose of study medication to the date of the first documentation of objective tumor progression or death on treatment due to any cause, whichever occured first (maximum 374 weeks)
Population: All participants who were enrolled and received at least 1 dose of study treatment, and had adequate baseline tumor assessment by either RECIST 1.1 or Cheson criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 16 | 9 | 18
Percentage of participants | 56.3 [33.2 to 76.9] | 66.7 [35.4 to 87.9] | 16.7 [5.8 to 39.2]

8. Secondary Outcome: Progression-Free Survival (PFS) Based on Investigator Assessement
Description: PFS was defined as the time from the date of first dose of study medication to the date of the first documentation of objective tumor progression (at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study [this includes the baseline sum if that is the smallest on study]). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered a sign of progression) or death on treatment due to any cause, whichever occured first. If tumor progression data included more than 1 date, the first date was used. The median PFS was estimated using Kaplan-Meier method.
Time Frame: From the date of first dose of study medication to the date of the first documentation of objective tumor progression or death on treatment due to any cause, whichever occurs first (maximum 444 weeks)
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 17 | 9 | 18
Months | NA [2.1 to NA] — Median PFS and upper limit of Confidence Interval not estimable due to insufficient number of participants with event. | NA [11.1 to NA] — Median PFS and upper limit of Confidence Interval not estimable due to insufficient number of participants with event. | 1.4 [1.1 to 4.9]

9. Secondary Outcome: Duration of Response (DR) Based on Investigator Assessement
Description: DR was defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. If tumor progression data included more than 1 date, the first date was used. CR: disappearance of all lesions; any pathological lymph nodes (target lesions [TLs]) or non-target lesions (non-TLs) must have reduction in short axis to <10 mm; normalization of tumor marker level for non-TLs; PR: >=30% decrease in sum of diameter of all TLs, taking as reference baseline sum of diameters; DR (in weeks) was calculated as (first date of PD or death - first date of CR or PR +1)/7. The median DR was estimated using Kaplan-Meier estimates.
Time Frame: From the first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first (maximum 374 weeks)
Population: Participants enrolled and treated who had baseline tumor assessment result and had confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 9 | 6 | 3
Weeks | NA [NA to NA] — Median DR and upper limit of Confidence Interval not estimable due to insufficient number of participants with event. | NA [30.1 to NA] — Median DR and upper limit of Confidence Interval not estimable due to insufficient number of participants with event. | NA [16.1 to NA] — Median DR and upper limit of Confidence Interval not estimable due to insufficient number of participants with event.

10. Secondary Outcome: Percentage of Participants Surviving at 6 Months and 1 Year
Description: The probability of survival at 6 months and 1 year, respectively, after the date of the first dose based on the Kaplan-Meier estimate.
Time Frame: At 6 months and 1 year after first dose
Population: Enrolled participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 17 | 9 | 18
Percentage of participants
  6 Months | 76.5 [48.8 to 90.4] | 100.0 [100.0 to 100.0] | 52.9 [27.6 to 73.0]
  1 Year | 70.6 [43.1 to 86.6] | 100.0 [100.0 to 100.0] | 52.9 [27.6 to 73.0]

11. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of first dose of study medication to the date of death due to any cause. OS (in months) was calculated as (date of death - date of first dose +1)/30.42. For participants still alive at the time of the analysis, for those who were lost to follow-up, and those who withdrew consent for additional follow up, the OS was censored on the last date that participants were known to be alive. Participants lacking data beyond the first dose had their OS censored at the date of first dose. The median OS was estimated using Kaplan-Meier method.
Time Frame: From the first dose of study treatment to the date of death due to any cause (maximum 444 weeks)
Population: Enrolled participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 17 | 9 | 18
Months | NA [7.5 to NA] — Median OS and upper limit of Confidence Interval not estimable due to insufficient number of participants with event. | NA [32.1 to NA] — Median OS and upper limit of Confidence Interval not estimable due to insufficient number of participants with event. | 12.6 [2.2 to 27.0]

12. Secondary Outcome: Steady-State Pre-dose Concentration (Ctrough) for Crizotinib on Day 1 of Cycles 2, 3 and 5
Description: Ctrough is defined as the drug concentration observed at the last planned timepoint prior to dosing. Steady state is defined as the participant receiving at least 90% of Crizotinib 500 mg daily dosing 14 days prior to the PK sample collection.
Time Frame: Predose within 1.2 hours before dosing on Day 1 of Cycles 2, 3 and 5
Population: Number of Participants Analyzed = participants who were enrolled and treated, had at least 1 PK blood sample collected, and were evaluable for steady-state Ctrough analysis. Number Analyzed = participants evaluable for this OM and had Ctrough data on the specific day.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 15 | 8 | 12
nanogram per milliliter (ng/mL)
  Cycle 2 Day 1: number analyzed (Participants) | 10 | 6 | 6
  Cycle 2 Day 1 | 270 (46.2) | 266 (42.0) | 233 (101)
  Cycle 3 Day 1: number analyzed (Participants) | 11 | 6 | 4
  Cycle 3 Day 1 | 316 (33.4) | 179 (92.1) | 187 (224)
  Cycle 5 Day 1: number analyzed (Participants) | 9 | 7 | 4
  Cycle 5 Day 1 | 244 (80.0) | 257 (35.1) | 347 (63.1)

13. Secondary Outcome: Steady-State Ctrough for PF-06260182 on Day 1 of Cycles 2, 3 and 5
Description: as for outcome 12
Time Frame: Predose within 1.2 hours before dosing on Day 1 of Cycles 2, 3 and 5
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 15 | 8 | 12
ng/mL
  Cycle 2 Day 1: number analyzed (Participants) | 12 | 7 | 10
  Cycle 2 Day 1 | 79.7 (64.6) | 68.2 (56.4) | 54.6 (123)
  Cycle 3 Day 1: number analyzed (Participants) | 12 | 6 | 7
  Cycle 3 Day 1 | 85.4 (88.2) | 41.7 (147) | 50.5 (566)
  Cycle 5 Day 1: number analyzed (Participants) | 9 | 7 | 5
  Cycle 5 Day 1 | 81.7 (96.8) | 71.9 (48.2) | 91.7 (68.7)

14. Secondary Outcome: Ctrough Ratios of PF-06260182 to Crizotinib on Day 1 of Cycles 2, 3 and 5
Description: Ctrough is defined as the drug concentration observed at the last planned timepoint prior to dosing. Steady state is defined as the participant receiving at least 90% of Crizotinib 500 mg daily dosing 14 days prior to the PK sample collection. The ratio is calculated as: (PF-06260182 concentration/464.33)/(Crizotinib concentration/450.34), where 464.33 is molecular weight for PF-06260182 and 450.33 is molecular weight for Crizotinib.
Time Frame: Predose within -1.2 hours before dosing on Day 1 of Cycles 2, 3 and 5
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 15 | 8 | 12
Ratio
  Cycle 2 Day 1: number analyzed (Participants) | 10 | 6 | 6
  Cycle 2 Day 1 | 0.323 (15.2) | 0.249 (25.0) | 0.190 (32.7)
  Cycle 3 Day 1: number analyzed (Participants) | 11 | 6 | 4
  Cycle 3 Day 1 | 0.314 (26.0) | 0.226 (41.4) | 0.126 (108)
  Cycle 5 Day 1: number analyzed (Participants) | 9 | 7 | 4
  Cycle 5 Day 1 | 0.326 (28.3) | 0.270 (27.7) | 0.243 (28.0)

15. Secondary Outcome: Number of Participants With ALK Genetic Events
Description: Number of participants with ALK translocation/fusion, amplification, mutation and overexpression at baseline assessed by technologies including fluorescence in-situ hybridization (FISH), immunohistochemistry (IHC), quantitative Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), ALK Fusion partners assessed by FISH or PCR; ALK gene amplification assessed by FISH or array Comparative Genomic Hybridization (aCGH), ALK Mutation assessed by PCR or direct sequencing were reported.
Time Frame: From Screening 28 Days Prior to Dosing Up to End of Treatment/Withdrawal (Maximum Up to Approximately 11 Years)
Population: The analysis planned to include all participant who had at least one dose of study treatment and at least one data of molecular profiling. Number Analyzed = participants who were enrolled and evaluable for this OM that had ALK genetic events at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 17 | 9 | 18
Participants
  ALK FISH | 2 | 9 | 12
  ALK Fusion Partner | 1 | 1 | 2
  ALK RT-PCR | 4 | 0 | 2
  ALK Gene Amplification | 0 | 0 | 3
  ALK IHC | 15 | 1 | 3
  ALK Mutation | 0 | 0 | 4

16. Secondary Outcome: Phosphorylation Status of ALK in the Tumor Samples From Surgery or Biopsy Pre and Post Treatment
Description: Tumor sample was planned to be provided to the designated central laboratory for retrospective confirmation of ALK phosphorylation status by a Pfizer designated central laboratory. The molecular profiling results were planned to include ALK fusion/translocation, mutations, amplification and overexpression.
Time Frame: From Screening 28 Days Prior to Dosing Up to End of Treatment/Withdrawal (Maximum Up to Approximately 11 Years)
Population: Analysis population included all participant who had at least one dose of study treatment and at least one data of molecular profiling at baseline and at end of treatment. Data were not collected due to that post-treatment tumor sample collection was optional per protocol and no participant had the post-treatment sample taken.
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment up to 28 days after the last dose of study treatment (maximum duration between first and last dose: 444 weeks)
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | ALCL Arm | IMT Arm | Other Tumors
All-Cause Mortality (participants affected / at risk) | 5/17 | 3/9 | 13/18
Serious Adverse Events (participants affected / at risk) | 8/17 | 4/9 | 7/18
Other Adverse Events (participants affected / at risk) | 16/17 | 9/9 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALCL Arm (N=17) | IMT Arm (N=9) | Other Tumors (N=18)
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 2 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALCL Arm (N=17) | IMT Arm (N=9) | Other Tumors (N=18)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 2
Lymph node pain (Blood and lymphatic system disorders) | 2 | 0 | 0
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 1 | 1
Myelosuppression (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 1
Blindness unilateral (Eye disorders) | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 2 | 0 | 0
Visual impairment (Eye disorders) | 8 | 4 | 5
Vitreous floaters (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 0 | 2
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 11 | 3 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 5 | 7
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 10 | 3 | 6
Asthenia (General disorders) | 7 | 0 | 2
Chest discomfort (General disorders) | 0 | 1 | 2
Chest pain (General disorders) | 2 | 0 | 1
Cyst (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 4 | 1 | 5
Gait disturbance (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 5 | 3 | 6
Pain (General disorders) | 1 | 0 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 10 | 1 | 2
Swelling face (General disorders) | 1 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Eyelid folliculitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 5 | 1 | 1
Klebsiella infection (Infections and infestations) | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 6 | 1 | 2
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Pelvic infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Paternal exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 9 | 4 | 5
Amylase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 4 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 4 | 2 | 0
Blood creatinine increased (Investigations) | 3 | 2 | 1
Blood folate decreased (Investigations) | 1 | 0 | 0
Blood glucose decreased (Investigations) | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 3 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Blood testosterone decreased (Investigations) | 1 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 2 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 1
Globulins decreased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 3 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 2 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 2 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 2 | 1 | 0
White blood cell count decreased (Investigations) | 5 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ageusia (Nervous system disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 6 | 1 | 2
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Petit mal epilepsy (Nervous system disorders) | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 1 | 2
Tremor (Nervous system disorders) | 1 | 1 | 0
Visual perseveration (Nervous system disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 2
Libido decreased (Psychiatric disorders) | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hair disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Abscess drainage (Surgical and medical procedures) | 0 | 0 | 1
Mole excision (Surgical and medical procedures) | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-08-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT01121588/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT01121588/SAP_001.pdf